CLINICAL TRIAL: NCT07280403
Title: Effect of a Low-carbohydrate Diet on Weight Loss in People Using the Injectable GLP-1 Agonist Semaglutide for Weight Loss: a Pilot Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: INQUIS Clinical Research (Industry)
Collaborators: Simply Good Foods USA, Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INQ-2411
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Weight Loss
Keywords: GLP-1 agonist; Semaglutide; Ozempic; Wegovy
MeSH Terms: conditions — Weight Loss | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: Randomized, open-label parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Carbohydrate (Experimental): Subjects randomized to the low-carbohydrate arm will be instructed on a reduced calorie diet (<1400 kcal/day) consisting of an average macronutrient distribution of 20% carbohydrate, 30% protein and 50% fat with a maximum intake of 40g/day of available (net) carbohydrates (approximately 65-75g total carbohydrates). To complement the provided low carbohydrate shakes and snacks, dietary counselling will focus on choosing sources of protein and non-starchy vegetables
  Interventions: Behavioral: Low Carbohydrate
- Low Fat (Active Comparator): Subjects randomized to the low-fat arm will be instructed on a reduced calorie diet (<1400 kcal/day) consisting of an average macronutrient distribution of 50% carbohydrate, 20% protein and 30% fat, with a maximum intake of 50g/day of fat. To complement the provided low fat shakes and snacks, dietary counselling will focus on choosing lean sources of protein and carbohydrates, while limiting high fat foods such as oils, nuts, full fat dairy, and fatty meats.
  Interventions: Behavioral: Low Fat

INTERVENTIONS:
Behavioral: Low Carbohydrate — Low carbohydrate diet
  Arms: Low Carbohydrate
Behavioral: Low Fat — Low fat diet
  Arms: Low Fat

SUMMARY:
The goal of this clinical trial is to determine the effect of a low carbohydrate higher protein diet, modelled after the Atkins program on weight loss, glycemic control, risk markers of cardiovascular disease and body composition in patients taking semaglutide.

Participants will:

* Be randomized to follow either a low carb, higher protein diet or a low fat diet for 3 months.
* Visit the clinic at week 2, 4, 8 and 12 to meet with a dietician, fill out a symptoms questionnaire and for bloodwork
* Complete 3-day food records 4 times over the 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years, inclusive
* Overweight or obese individuals with a BMI ≥26 kg/m²
* Non-pregnant, non-lactating individuals who are not planning on becoming pregnant during the trial and are using an effective method of contraception, as outlined: (a) Complete abstinence from intercourse two weeks prior to administration of the study product, and throughout the clinical trial. Participants utilizing this method must agree to use 2 alternate methods of contraception (see d) if they should become sexually active and will be queried on whether they have been abstinent at each study visit. b) Has a male sexual partner who is surgically sterilized prior to the Screening Visit and is the only male sexual partner for that Participant; c) Sexual partner(s) is/are exclusively female; d) Use of two acceptable methods of contraception, such as a spermicide, mechanical barrier (e.g. male condom, female diaphragm), tubal ligation, contraceptive pill, intrauterine device (IUD) or contraceptive implant. The Participant must be using these methods for at least 1 week prior to the screening visit and throughout their participation in the trial.
* Started semaglutide injections for weight loss 14 to 35 days prior to screening, inclusive, are tolerating it and are willing to continue taking it
* HbA1c ≤7.5%
* Not taking any hypoglycemic agent, apart from a semaglutide
* Systolic blood pressure <160 mmHg and diastolic blood pressure <100 mmHg
* Serum creatinine <180 mmol/L (<2.1 mg/dL)
* Serum triglycerides <9 mmol/L (<800 mg/dL)
* ALT or AST <3 times the upper limit of normal
* Untreated LDL-cholesterol <5.00 mmol/l (<193 mg/dL)
* No major illness, trauma or surgery requiring hospitalization within 3mo of the screening visit
* Ability to understand the study procedures and willing to provide informed consent to participate in the study
* Subjects must be eligible to receive income in Canada and be covered by a health insurance plan such as OHIP
* Subjects are willing to sign the informed consent prior to any procedures conducted

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* High alcohol consumption (>14 standard drinks per week or >4 standard drinks per day for males; and > 7 standard drinks per week or >3 standard drinks per day for females), with 1 standard drink defined as containing approximately 14g of pure alcohol. Examples of 1 standard drink include: 12 oz of regular beer (approx. 5% alcohol), 5 oz of wine (approx. 12% alcohol) or 1.5 oz of distilled spirits (approx. 40% alcohol)
* Individuals with a history of bariatric surgery, gastrointestinal disease, any other medical conditions or use of supplements or medications that increase risk to the subject or others or may affect the results, as judged by the Principal Investigator
* Unwillingness or inability to comply with the experimental procedures and to follow INQUIS safety guidelines
* Known intolerance, sensitivity, or allergy to any ingredients in the study test products
* Subject is currently participating or recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement, or lifestyle modification

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Body weight | 12 weeks
  Percentage change from baseline of body weight

SECONDARY OUTCOMES:
BMI | 12 weeks
  Change from baseline of BMI
Fat Mass | 12 weeks
  Change from baseline of Fat Mass
Fasting plasma glucose | 12 weeks
  Change from baseline of fasting plasma glucose
Fat-free mass | 12 weeks
  Change from baseline of Fat-Free Mass
Skeletal Muscle Mass | 12 weeks
  Change from baseline of Skeletal Muscle Mass
Fasting serum insulin | 12 weeks
  Change from baseline of fasting serum insulin
Insulin sensitivity index | 12 weeks
  Change from baseline of HOMA-IR

CONTACTS AND LOCATIONS:
Overall Officials: Janice Campbell, Study Director — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Permission has not been sought to do so. Not shared to protect personal health information and participant identity.